CLINICAL TRIAL: NCT04081818
Title: A Study on the Effects of Nutritious Mushrooms in Adults With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Responsible Party: Principal Investigator, Andriana C Kaliora, Assistant Professor in Foods and Human Nutrition, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Nutritious_Mushrooms_61100
Record Dates: First submitted 2019-06-20; First posted 2019-09-09 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Nutritious Mushrooms) (Active Comparator)
  Interventions: Other: Nutritious Mushrooms
- Control group (No Intervention)

INTERVENTIONS:
Other: Nutritious Mushrooms — The Intervention group will consume antioxidant rich and Vitamin D2-enhanced mushrooms as a snack daily for 3 months.
  Arms: Intervention group (Nutritious Mushrooms)

SUMMARY:
Obesity, characterized by an increase in body weight that results in excessive fat accumulation, is a global health problem. Recently, it has also been shown that obesity is associated with low-grade chronic systemic inflammation in adipose tissue. This condition is mediated by activation of the innate immune system in adipose tissue that promotes inflammation and oxidative stress and triggers a systemic acute-phase response.

Previous research points towards the potential of phytochemicals in food as part of nutritional strategies for the prevention of obesity and associated inflammation, as well as, increase in insulin sensitivity in diabetic patients.

In addition, there is strong evidence that obesity is inversely associated with vitamin D levels. The major cause of vitamin D deficiency in humans is the lack of adequate sun exposure. Unfortunately, very few foods, i.e. mushrooms, naturally contain vitamin D and foods that are fortified with vitamin D are inadequate to satisfy vitamin D requirements.

The last decade, mushrooms have attracted the research interest as functional foods with desirable health benefits in several metabolic disorders without the side effects of pharmacological treatment. Edible mushrooms are highly nutritious and exhibit beneficial effects on several inflammatory diseases such as cancer, heart disease, diabetes,, high blood pressure.

Thus, the purpose of this study is to determine the effects of nutritious mushrooms in adults with Metabolic Syndrome. More specifically, 100 participants will be allocated to two groups, namely intervention group (N=50) and control group (N=50). Vitamin D2-enhanced mushrooms by UV-B will be provided as a snack to the intervention group, whereas the control group will not consume the snack. The intervention will last 3 months.The effects of the intervention will be evaluated via clinical and laboratory markers. Personal and family history, anthropometric, demographic data, body composition, dietary habits, physical activity and smoking status will be assessed pre- and post- intervention. Biochemical profile, oxidative stress and inflammation, as well as metabolomic profiles will be assessed in blood samples pre- and post- intervention. Both groups will receive standard nutritional counselling throughout the intervention and will be encouraged to report any adverse effects they may experience during the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 30 years < Age < 65 years
* BMI > 25 kg/ m2
* Metabolic Syndrome

Exclusion Criteria:

* Hepatotoxic Medication
* Diabetes Mellitus
* Dysthyroidism, hypopituitarism, Cushing syndrome / disease
* Pregnancy, lactation
* Psychiatric or mental disorder
* Any use of antioxidant-phytochemical rich supplement, vitamin D supplement, nti-, pre- or pro-biotics within 3 months pre-intervention

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity change pre- and post- intervention in each arm, measuring fasting blood sugar levels. | 3 months

SECONDARY OUTCOMES:
Vitamin D2 levels change pre- and post- intervention in each arm | 3 months
Anthropometric measures change pre- and post- intervention in each arm | 3 months
Biochemical markers change pre- and post- intervention in each arm | 3 months
Inflammation and oxidative stress markers change pre- and post- intervention in each arm | 3 months
Quality of life change pre- and post- intervention in each arm | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Andriana Kaliora, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marseglia L, Manti S, D'Angelo G, Nicotera A, Parisi E, Di Rosa G, Gitto E, Arrigo T. Oxidative stress in obesity: a critical component in human diseases. Int J Mol Sci. 2014 Dec 26;16(1):378-400. doi: 10.3390/ijms16010378. PMID 25548896
- [Background] Cardwell G, Bornman JF, James AP, Black LJ. A Review of Mushrooms as a Potential Source of Dietary Vitamin D. Nutrients. 2018 Oct 13;10(10):1498. doi: 10.3390/nu10101498. PMID 30322118
- [Background] Abdali D, Samson SE, Grover AK. How effective are antioxidant supplements in obesity and diabetes? Med Princ Pract. 2015;24(3):201-15. doi: 10.1159/000375305. Epub 2015 Mar 14. PMID 25791371
- [Background] Duggan C, de Dieu Tapsoba J, Mason C, Imayama I, Korde L, Wang CY, McTiernan A. Effect of Vitamin D3 Supplementation in Combination with Weight Loss on Inflammatory Biomarkers in Postmenopausal Women: A Randomized Controlled Trial. Cancer Prev Res (Phila). 2015 Jul;8(7):628-35. doi: 10.1158/1940-6207.CAPR-14-0449. Epub 2015 Apr 23. PMID 25908506
- [Background] Norman PE, Powell JT. Vitamin D and cardiovascular disease. Circ Res. 2014 Jan 17;114(2):379-93. doi: 10.1161/CIRCRESAHA.113.301241. PMID 24436433
- [Background] Holick MF, Chen TC. Vitamin D deficiency: a worldwide problem with health consequences. Am J Clin Nutr. 2008 Apr;87(4):1080S-6S. doi: 10.1093/ajcn/87.4.1080S. PMID 18400738
- [Background] Mutt SJ, Hypponen E, Saarnio J, Jarvelin MR, Herzig KH. Vitamin D and adipose tissue-more than storage. Front Physiol. 2014 Jun 24;5:228. doi: 10.3389/fphys.2014.00228. eCollection 2014. PMID 25009502
- [Background] Urbain P, Singler F, Ihorst G, Biesalski HK, Bertz H. Bioavailability of vitamin D(2) from UV-B-irradiated button mushrooms in healthy adults deficient in serum 25-hydroxyvitamin D: a randomized controlled trial. Eur J Clin Nutr. 2011 Aug;65(8):965-71. doi: 10.1038/ejcn.2011.53. Epub 2011 May 4. PMID 21540874
- [Background] El Khoury D, Cuda C, Luhovyy BL, Anderson GH. Beta glucan: health benefits in obesity and metabolic syndrome. J Nutr Metab. 2012;2012:851362. doi: 10.1155/2012/851362. Epub 2011 Dec 11. PMID 22187640
- [Background] Ganesan K, Xu B. Anti-Obesity Effects of Medicinal and Edible Mushrooms. Molecules. 2018 Nov 5;23(11):2880. doi: 10.3390/molecules23112880. PMID 30400600